CLINICAL TRIAL: NCT06188429
Title: Peripheral Blood VA/TREM2 Levels and Their Correlation Analysis With the Development and Autistic Symptoms in Children With ASD
Acronym: PBVTLCAASD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hua Wei (Other)
Responsible Party: Sponsor-Investigator, Hua Wei, Dr, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Other Study IDs: (2023) Lund Review No.452
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: ASD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group: Children with ASD
  Interventions: Diagnostic Test: DSM-5
- Control Group: Normal Children
  Interventions: Diagnostic Test: DSM-5

INTERVENTIONS:
Diagnostic Test: DSM-5 — Using DSM-5 for diagnostic testing of the children in the study group.

SUMMARY:
Autism Spectrum Disorder (ASD) is a neurodevelopmental disorder characterized by social impairment, repetitive behaviors, and narrow interests. With advancements in diagnostic techniques, the prevalence of ASD has been increasing annually. However, due to its complex and diverse etiology, there is no definitive consensus on the pathogenic mechanism of ASD. Numerous studies indicate that genetics, environment, and other factors play crucial roles in the onset of ASD.

Vitamin A (VA) exerts its effects in the body through its active metabolite, retinoic acid (RA), which regulates the transcriptional activity and expression of downstream genes by binding to retinoic acid receptors (RARs/RXRs). Triggering Receptor Expressed on Myeloid Cells 2 (TREM2) is an immunoglobulin-like receptor present on microglial cells, with functions including inhibiting the production of inflammatory factors and engulfing apoptotic neurons. Recent foreign studies show a significant decrease in TREM2 levels in the brain tissue of ASD patients. However, there is limited research on the relationship between TREM2 and ASD.

In our previous animal experiments, we observed a reduction in TREM2 in the prefrontal cortex of the brain in ASD model rats. Administering overexpressed TREM2 improved autism-like behavior in ASD model rats, and supplementing RA upregulated the expression of RA-RARα and TREM2, modulated microglial cell activation, and improved autism-like behavior in rats. Therefore, we believe that the RA/RARα pathway regulates the TREM-2 signaling pathway, mediating changes in microglial cells, and TREM2 may be involved in the pathogenesis of ASD.

Soluble TREM2 (sTREM2) is formed by the extracellular domain shedding of TREM2 under the action of ADAM protease. Research indicates that the expression of sTREM2 can be detected in cerebrospinal fluid and plasma. However, the connection between VA, sTREM2 levels, and the behavioral and developmental levels of children with ASD remains unclear and requires further clinical research to validate. This will help deepen our understanding of TREM2 expression in ASD, its potential biological functions, and the role of RA.

ELIGIBILITY:
Inclusion Criteria:

* The Children's Health Department (Health Management Department) of Chongqing Medical University Affiliated Children's Hospital is recruiting 50 typical children and 50 children with ASD. Disease diagnosis will be conducted by professional doctors, and ASD diagnosis must comply with the DSM-5 diagnostic criteria.

Exclusion Criteria:

* Patients or their family members unable to cooperate with blood collection for testing are excluded. Exclusion criteria also involve a history of other neurological disorders, chromosomal diseases, genetic metabolic disorders, and other significant physical illnesses such as auditory or visual impairments, epilepsy, phenylketonuria, tuberous sclerosis, neurofibromatosis, severe head trauma, autoimmune diseases, and disorders related to the endocrine, cardiovascular, pulmonary, hepatic, or renal systems. Patients' legal guardians refusing to participate in the project are also excluded.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The Children's Health Department (Health Management Department) of Chongqing Medical University Affiliated Children's Hospital is recruiting 50 children with ASD and 50 typical children, aged between 3 and 8 years old. ASD diagnosis must comply with the DSM-5 diagnostic criteria.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Blood VA/sTREM2 level | 3 months
  Using an ELISA assay kit to detect the serum sTREM2 levels and employing high-performance liquid chromatography (HPLC) to measure the Vitamin A content in peripheral blood.

SECONDARY OUTCOMES:
Autistic Symptoms | 1 week
  Using the ADOS (Autism Diagnostic Observation Schedule) scale to analyze the severity of autism symptoms in autistic children.

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing Medical University Affiliated Children's Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No